CLINICAL TRIAL: NCT03556488
Title: Prognostic Role of Ultrasonographic Air Bronchogram in the Management of Community Acquired Pneumoniae in Children
Brief Title: Ultrasonographic Air Bronchogram in Pediatric CAP
Acronym: USINCHILD
Status: Recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Riccardo Inchingolo, Physician and clinical researcher, Catholic University of the Sacred Heart
Other Study IDs: 13528/18
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pneumonia; Pediatric Infectious Disorder
Keywords: Chest ultrasound; Pediatric community acquired pneumonia; Air bronchogram
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric CAP: Patients with a clinical diagnosis of CAP and radiographic evidence of lung consolidation, hospitalized in the Pediatric Unit.
  Interventions: Diagnostic Test: US air bronchogram score

INTERVENTIONS:
Diagnostic Test: US air bronchogram score — On ultrasonographic examination, lung consolidation is defined as a subpleural echo-poor region or one with tissue- like echotexture, depending on the extent of air loss and fluid predominance, which is clearly different from the normal pattern.
  The air bronchogram is characterized as: absent, static, dynamic, dynamic with areas of lung recruitment.

SUMMARY:
This study evaluates the prognostic role of the change of arborescent air bronchogram, a typical ultrasonographic finding of lung consolidation due to pneumonia, in the management of pediatric CAP.

DETAILED DESCRIPTION:
This is a single-center prospective study to evaluate the prognostic role of the change of arborescent air bronchogram, a typical ultrasonographic finding of lung consolidation due to pneumonia, in the management of CAP in terms of: 1) impact on rate of uncomplicated respiratory infections [rate of uncomplicated CAP], 2) relationship to the time of resolution of clinical signs [time to resolution of fever], 3) change of antibiotic therapy not guided by microbiological examinations and, 4) length of hospitalization.

At admission, the Pediatric will evaluate clinical signs of respiratory distress, request microbiologic tests (nasopharyngeal swab specimens and pneumococcal urinary antigen) to detect causative pathogens of CAP, and laboratory tests (complete blood cell count, acute-phase reactants C-reactive protein). Finally, all children will undergo chest radiography (CXR). If CXR should be performed before the admission to Pediatric Unit, the radiological exam will be not repeated.

Ultrasonographic evaluation will be performed by Pulmonologists. The first examination will be performed within 12 hours from admission. The Pulmonologists will be blind to clinical and radiological data.

In order to characterize the lung consolidation, a grading system based on the presence and the features of air bronchogram [static, dynamic, dynamic with areas of lung recruitment] will be adopted. The operator will collect and store images and videos (10seconds), these findings will be reviewed by an expert Clinician in chest US blind to other data.

After 48h from the admission, all children will undergo follow-up laboratory tests and lung US.

In case of clinical deterioration, children will undergo further ultrasonographic evaluations according pediatric indications.

Finally, all children will undergo lung US after 7 ± 2 days from discharge.

ELIGIBILITY:
Inclusion Criteria:

* Suspected CAP
* Age from 1 to 16 years old
* Admission to Pediatric Unit
* Radiographic evidence of lung consolidation
* Written informed consent from parents

Exclusion Criteria:

* Gestational age < 36 weeks
* Previous diagnosis of cystic fibrosis
* Congenital pulmonary disease.
* Refusal to participate.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a clinical diagnosis of CAP and radiographic evidence of lung consolidation.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of uncomplicated CAP | 48 hours
  Impact on rate of uncomplicated respiratory infections
Time to resolution of fever | Through study completion, an average of 7 days.
  Relationship to the time of resolution of clinical signs
Change of antibiotic therapy | 48 hours
  Change of antibiotic therapy not guided by microbiological examinations
Length of hospitalization | Through study completion, an average of 10 days.
  Length of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Luca Richeldi, Prof,MD,PhD, Study Director — Fondazione Policlinico Universitario A. Gemelli, IRCCS; Riccardo Inchingolo, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Azienda Sanitaria Universitaria Integrata di Trieste - Ospedale di Cattinara, Trieste

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Inchingolo R, Copetti R, Smargiassi A, Gerardi RE, Conte EG, Corbo GM, Gatto A, Pierandrei C, Capossela L, Lazzareschi I, Valentini P, Demi L. Air bronchogram integrated lung ultrasound score to monitor community-acquired pneumonia in a pilot pediatric population. J Ultrasound. 2021 Jun;24(2):191-200. doi: 10.1007/s40477-020-00547-7. Epub 2021 Jan 6. PMID 33409860